CLINICAL TRIAL: NCT01229085
Title: CLINICAL ASSESSMENT OF THE EFFECTIVENESS OF ASSOCIATION MONETASONE FUROATE 0.1% SALICYLIC ACID AND 5% FOR SUBMISSION OF OINTMENT TOPICAL DERMATOLOGICAL USE OF LABORATORY Glenmark Pharmaceuticals Ltd, IN PATIENTS WITH PSORIASIS.
Brief Title: Efficacy Study of the Combination Mometasone + Salicylic Acid in Patients With Psoriasis
Acronym: Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SALMOGLEN20906
Record Dates: First submitted 2008-02-08; First posted 2010-10-27 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2008-02

CONDITIONS: Psoriasis
Keywords: Psoriasis, mometasone, salicylic acid.
MeSH Terms: conditions — Psoriasis | interventions — Salicylic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Test (Experimental): mometasone 0,1% + salicylic acid 5%
  Interventions: Drug: memotasone + salicylic acid

INTERVENTIONS:
Drug: memotasone + salicylic acid — mometasone 0,1% + salicylic acid 5%.

SUMMARY:
To evaluate the efficacy of the combination of mometasone furoate 0.1% and Salicylic Acid 5% in patients of both sexes who presented clinical symptoms of psoriasis of mild to moderate.

DETAILED DESCRIPTION:
Phase III clinical trial, systematic sampling, open-label study that evaluated the efficacy of the combination of mometasone furoate 0.1% and 5% salicylic acid in 71 patients with lesions of mild to moderate psoriasis treated for up to 45 days or less than this, at the discretion of the investigator. The results were statistically analyzed and investigational data and their conclusions are referred to in this report.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes, regardless of color or social class;
* Age 18 or older, with good mental health;
* Psoriasis patients with mild to moderate;
* Patients who agreed to participate and signed the
* Clarified (appendix);
* Patients who agreed to return for follow-up visits.

Exclusion Criteria:

* Patients who were making use of biologics, corticosteroids or nonsteroidal anti-inflammatory and non-steroid, or who made use of these topical medications until 15 days before inclusion or 30 days before inclusion when the administration was orally;
* Patients who were exposed to the sun 15 days before the study began or during the course of the same;
* Patients who were making use of acetaminophen;
* Patients who did not agree to the terms described in the IC informed consent, - Patients who also had psoriatic plaques of skin disorders caused by fungi or bacteria and they were making use of antibiotic or antifungal;
* Lions and other types of skin damage that was not psoriasis;
* Pregnant and nursing women;
* Patients using oral anticoagulants.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To assess the safety in use as primary end point and end point as effectively isolated secondary association in patients with plaque psoriasis of mild to moderate. | 45 days of treatment.
  Patients will visit the center at weeks 0, 1, 2, 4 and 6 totaling 45 days. Parameters will be evaluated for erythema, plaque size, scaling, itching, thickness of the lesion as well as recording and analysis of adverse effects from treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clinica Pesquisa e Desenvolvimento Ltda., Valinhos, São Paulo, Brazil